CLINICAL TRIAL: NCT06868290
Title: A Phase 2, Randomized, Open-label, Controlled Study to Evaluate the Efficacy and Safety of Rapcabtagene Autoleucel Versus Comparator in Participants With Severe Active Granulomatosis With Polyangiitis (GPA) or Microscopic Polyangiitis (MPA)
Brief Title: Phase 2 Study Evaluating Rapcabtagene Autoleucel in Participants With Severe Active GPA or MPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYTB323I12201
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: ANCA Associated Vasculitis (AAV)
Keywords: Chimeric Antigen Receptor-T (CAR-T); rapcabtagene autoleucel; anti-neutrophil cytoplasmic antibody (ANCA); ANCA-associated vasculitis/vasculitides (AAV); Granulomatosis with Polyangiitis (GPA); Microscopic Polyangiitis (MPA)
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Glucocorticoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study investigator and the participant will be unblinded to the study treatment. A blinded assessor will perform the efficacy assessments to minimize bias in data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapcabtagene autoleucel (Experimental): Single infusion of rapcabtagene autoleucel (YTB323) and concomitant glucocorticoids as per protocol
  Interventions: Biological: Rapcabtagene autoleucel; Drug: Glucocorticoids
- Active comparator (Active Comparator): Comparator and concomitant glucocorticoids as per protocol
  Interventions: Other: Active Comparator; Drug: Glucocorticoids

INTERVENTIONS:
Biological: Rapcabtagene autoleucel — Single infusion of rapcabtagene autoleucel
  Arms: Rapcabtagene autoleucel
Other: Active Comparator — Active comparator option as per protocol
  Arms: Active comparator
Drug: Glucocorticoids — Concomitant glucocorticoids as per protocol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rapcabtagene autoleucel versus comparator in participants with severe active Granulomatosis with Polyangiitis (GPA) or Microscopic Polyangiitis (MPA)

DETAILED DESCRIPTION:
This is a Phase 2, randomized, assessor-blinded active controlled study. This study comprises two cohorts:

* A lead-in cohort enrolling participants to receive rapcabtagene autoleucel
* A randomized cohort with participants receiving either rapcabtagene autoleucel or comparator.

After end of study (EOS), participants who received rapcabtagene autoleucel infusion will enter a long-term follow-up (LTFU) period lasting up to 15 years after rapcabtagene autoleucel infusion. This LTFU will be described in a separate study protocol.

ELIGIBILITY:
Key inclusion criteria:

1. Men and women, aged ≥18 and ≤ 75 years with a diagnosis of GPA or MPA according to the American College of Rheumatology/ European League Against Rheumatism 2022 (ACR/EULAR 2022) classification criteria
2. Positive test for ANCA-autoantibodies
3. GPA and MPA participants with severe active disease

Key exclusion criteria:

1. Any condition that could prevent a complete washout of medications or could otherwise make the participant ineligible for anti-CD19 CAR-T therapy and further participation in the study
2. Hypersensitivity and/or contraindications to any product to be given to the participant as part of the study protocol
3. Other systemic autoimmune diseases requiring therapy
4. Any medical conditions that are not related to GPA/MPA that would jeopardize the ability of the participant to tolerate CD19 CAR-T cell therapy
5. Inadequate organ function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2029-06-07 (Estimated); Study Completion 2030-05-24 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From randomization until the occurrence of an EFS event, up to approx. 4 years after randomization
  Event-free survival (EFS) defined as the time from Randomization to the first occurrence of as per protocol defined events.

SECONDARY OUTCOMES:
Percentage of patients achieving complete remission | Up to Week 13
  Complete remission is defined by Birmingham Vasculitis Activity Score version 3 (BVASv3)
Adjusted annual cumulative GC dose between Randomization and analysis cutoff date | From randomization until the occurrence of an EFS event, up to approx. 4 years after randomization
  The adjusted annual cumulative glucocorticoid dose refers to the total amount of glucocorticoids administered to a patient over the course of a year, adjusted for any changes in dosage, and measured up to the defined week of treatment as per protocol.
ANCA seronegativity and sustaining ANCA seronegativity until the analysis cutoff date | From randomization until the occurrence of an EFS event, up to approx. 4 years after randomization
  ANCA seronegativity means that the patient tests negative for ANCA antibodies.
Change from baseline in estimated glomerular filtration rate (eGFR) at Week 39 | Up to Week 39
  Change from baseline in estimated glomerular filtration rate (eGFR) at Week 39.
Change from baseline in symptoms of GPA/ MPA using the AAV-PRO at Week 39 | Up to Week 39
  Change from baseline in symptoms of GPA/ MPA using the AAV-PRO at Week 39.
Change from baseline in Patient- Reported Outcome Measurement Information System (PROMIS)- Fatigue 7a at Week 91. | Up to Week 91
  Change from baseline in PROMIS- Fatigue 7a at Week 91.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (8):
  - University Of Colorado, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Oregon Health Sciences University, Portland, Oregon
  - Houston Methodist Hospital, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
- Japan (9):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
- United Kingdom (2):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided are anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com